CLINICAL TRIAL: NCT06719063
Title: Effect of Immersive Virtual Reality With Multisensory Stimulation on the Functional Impact of Hemineglect Secondary to a Right-Sided Stroke: A Single Case Experimental Design (SCED) Study
Brief Title: Effect of Immersive Virtual Reality With Multisensory Stimulation on the Functional Impact of Hemineglect Secondary to a Right-Sided Stroke
Acronym: NEGLISENS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital La Musse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-A01439-38
Record Dates: First submitted 2024-11-27; First posted 2024-12-05 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2024-11

CONDITIONS: Stroke; Hemineglect; Neuropsychology; Virtual Reality; Rehabilitation; Immersion
Keywords: stroke; hemineglect; neuropsychology; virtual reality; rehabilitation; multisensory; immersion
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): The evaluation sessions aim to measure the impact of hemineglect on autonomy. This measurement will be conducted using the Catherine Bergego Scale, which will be completed by both the patient and the occupational therapist. Evaluation sessions will last approximately 45 minutes and will take place once a week for 10 to 12 weeks.
  After 3 to 5 weeks of evaluations (Phase A: baseline), the patient will participate in three weekly rehabilitation sessions, each lasting 45 minutes, over a 5-week period (Phase B: therapy). These sessions will be individual and conducted by an occupational therapist. Each session will follow a similar structure: review of the previous session, explanation of the current session, a 15-minute multisensory experience using virtual reality, and a final review focusing particularly on tolerance.
  A multisensory experience has been specifically designed for the rehabilitation protocol. The experience consists of two 360° nature-themed films. Throughout the experie
  Interventions: Other: Multisensory Virtual Reality

INTERVENTIONS:
Other: Multisensory Virtual Reality — The VirtySens® multisensory travel capsule is an immersive virtual reality technique. This total immersion occurs through the simultaneous stimulation of four of the five senses.
  Session duration: 45 minutes, with 15 minutes dedicated to the protocol administration. The remaining 30 minutes will be used to welcome the patient, explain the content of the session, and review the session's outcome, particularly to assess tolerance (Simulator Sickness Questionnaire (SSQ) completed at the start of each week after the first VirtySens® session). The sessions will take place in the morning to prevent the session from being disrupted by fatigue related to the rehabilitation day.

SUMMARY:
A stroke is a common and potentially serious condition that affects 130,000 people each year in France. It is the second leading cause of major cognitive disorders after Alzheimer's disease.

Hemineglect is a frequently observed cognitive impairment following a stroke. The individual becomes unable to orient themselves or respond to stimuli appearing in the contralesional hemispace. Hemineglect occurs in approximately 25-30% of stroke patients, with the right hemisphere being affected in 90% of cases.

Despite potential spontaneous recovery within the first 2 to 3 months post-stroke, neglect tends to persist chronically. One-third of patients suffer from long-term neglect. The condition is more severe after a right-sided lesion. The functional impact is significant, particularly when considering the anosognosia and anosodiaphoria often associated with it. Rehabilitation stays are longer for patients with neglect, and autonomy in daily activities is reduced. Neglect leads to poorer functional outcomes after a stroke, making it a critical factor to address in a patient's rehabilitation program.

The goal of rehabilitation is to reduce impairments, improve activity limitations and participation restrictions secondary to hemineglect, and achieve functional progress beyond what is possible through spontaneous recovery. Since no single rehabilitation method for neglect is superior to another, it is currently recommended to combine multiple approaches.

The top-down approach is based on intention and conscious effort. This technique is among the first used for neglect rehabilitation and remains widely used today. The goal is to help the patient become aware of their neglectful behavior.

The bottom-up approach relies on more automatic mechanisms of action and aims to modulate the spatial reference system through passive sensory manipulations or visuomotor adaptation.

The use of virtual reality in stroke rehabilitation promotes plasticity and neural reorganization. In the field of hemineglect, several studies have examined the effects of virtual reality using top-down and/or bottom-up approaches and have shown significant functional improvements. In the case of multisensory stimulation, delivering different stimuli to the same side of space and at the same time increases neuronal activity, leading to a stronger clinical response than unisensory stimulation.

The VirtySens® multisensory travel capsule is an immersive virtual reality technique. This total immersion is achieved through the simultaneous stimulation of four out of the five senses. Firstly, vision and hearing are stimulated by a virtual reality headset that projects high-definition films. Smell is activated through the release of micro-droplets of fragrances synchronized with the imagery. Finally, touch is stimulated by warm and cold airflows that enhance the various scenes presented.

The investigators emit the hypothesis that the VirtySens® capsule, immersive virtual reality combining multisensory stimulation via four of the five senses and training in visual scanning, introduced in rehabilitation, allows to significantly reduce the functional impact of hemineglect in the adult victim of a right cerebral infarction dating less than 3 months.

To respond to these research objectives, the investigators will carry out a pilot study in Single Case Experimental Design (SCED). The experimentation will take place in mainland France within La Musse hospital. The recruitment of 3 subjects will be necessary for the realization of this study.

The study will consist of repeated evaluation and rehabilitation sessions. Evaluations will be conducted at La Musse Hospital by an occupational therapist. The purpose of the evaluation sessions is to measure the impact of hemineglect on autonomy. This measurement will be performed using the Catherine Bergego Scale, which will be completed by both the patient and the occupational therapist. Evaluation sessions will last approximately 45 minutes and will take place once a week for 10 to 12 weeks.

After 3 to 5 weeks of evaluations, the patient will participate in three weekly rehabilitation sessions, each lasting 45 minutes, over a 5-week period. These sessions will be individual and conducted by an occupational therapist. Each session will follow a similar structure: review of the previous session, explanation of the current session, a 15-minute multisensory experience using virtual reality, followed by a review of the session, particularly focusing on tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 18 years
* Diagnosis of first ischemic right stroke established by a neurologist using clinical examination and brain imaging (CT scan or MRI)
* Stroke occurring less than 3 months ago
* Presence of left hemineglect, diagnosed using the Neglect Assessment Battery (NAB)
* Normal vision or corrected to normal
* Patient affiliated with the social security system

Exclusion Criteria:

* History of neurological or psychiatric illness
* Epilepsy
* Craniotomy
* Limited range of cervical motion due to orthopedic disorders
* Moderate or severe deafness (hearing loss of 40 dB in one ear, as measured by tonal audiometry)
* Anosmia (loss of smell)
* Asthmatic disease
* Pregnant women or women suspected of being pregnant
* Breastfeeding women
* Severe neurocognitive disorders with an MMSE score < 21
* Patient under legal protection measures
* Minor patient
* Patient enrolled in another research protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
The impact of hemineglect on autonomy | From study enrollment, up to 12 weeks, every 7 days
  The evaluation sessions aim to measure the impact of hemineglect on autonomy. This measurement will be conducted using the Catherine Bergego Scale, which will be completed by both the patient and the occupational therapist. This scale is scored from 0 to 30 points; the higher the score, the more severe the behavioural neglect.

SECONDARY OUTCOMES:
The measurement of anosognosia or awareness of hemineglect | From study enrollment, up to 12 weeks, every 7 days
  The measurement of anosognosia or awareness of hemineglect in an ecological setting, using the Catherine Bergego Scale. This scale is scored from 0 to 30 points; the higher the score, the more severe the behavioural neglect.
The measurement of tolerance to immersive virtual reality | From study enrollment, up to 12 weeks, every 7 days
  The measurement of tolerance to immersive virtual reality, combining multisensory stimulation through four of the five senses and visual scanning training, introduced in rehabilitation, using the Simulator Sickness Questionnaire.
  This scale is scored from 0 to 48 points, the higher the score, the greater the cybermalaise.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital La Musse, Saint-Sébastien-de-Morsent, France

IPD SHARING:
Plan to Share IPD: Undecided